CLINICAL TRIAL: NCT00023868
Title: A Randomized Phase I/III Study Of Systematic Chemotherapy With Or Without Hepatic Chemoembolization For Liver-Dominant Metastatic Adenocarcinoma Of The Colon And Rectum
Brief Title: Combination Chemotherapy With or Without Chemoembolization in Treating Patients With Colorectal Cancer Metastatic to the Liver (6655)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: redesign
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068871; ACRIN-6655 (Other: American College of Radiology Imaging Network); U01CA079778 (NIH); U01CA080098 (NIH)
Record Dates: First submitted 2001-09-13; First posted 2003-06-17 (Estimated); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Cisplatin; Doxorubicin; Fluorouracil; Irinotecan; Leucovorin; Mitomycin

INTERVENTIONS:
Drug: FOLFIRI regimen
Drug: cisplatin
Drug: doxorubicin hydrochloride
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium
Drug: mitomycin C

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan, fluorouracil, and leucovorin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping the cells from dividing. Chemoembolization kills tumor cells by blocking the blood flow to the tumor and keeping chemotherapy drugs near the tumor. It is not yet known if chemoembolization is more effective than standard chemotherapy in treating metastatic cancer.

PURPOSE: This phase I trial and randomized phase III trial is studying the effectiveness of chemoembolization in treating patients who have colorectal cancer metastatic to the liver.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the survival of patients with liver-dominant metastatic colorectal adenocarcinoma treated with irinotecan, fluorouracil, and leucovorin calcium with or without hepatic chemoembolization.
* Compare response in the liver, time to hepatic tumor progression, and time to extrahepatic tumor progression in patients treated with these regimens.
* Compare the possible treatment differences with respect to morbidity, toxic effects of chemoembolization, toxic effects of chemotherapy, and death from cancer-related complications in these patients.

OUTLINE: This is a phase I dose-escalation study followed by a phase III randomized, multicenter study. (Phase I closed as of 10/14/02.)

* Phase I: Patients in phase I are sequentially enrolled to 1 of 3 treatment regimens. (Phase I closed as of 10/14/02.)

  * Regimen A: Patients receive irinotecan IV over 60-90 minutes, leucovorin calcium IV, and fluorouracil IV over 10 minutes on days 1, 8, 15, and 22. Patients undergo hepatic embolization with embolic suspension only on day 36.
  * Regimen B: Patients receive chemotherapy as in regimen A. Patients undergo hepatic chemoembolization with lower-dose cisplatin, doxorubicin, and mitomycin on day 36.
  * Regimen C: Patients receive chemotherapy as in regimen A. Patients undergo hepatic chemoembolization with higher-dose cisplatin, doxorubicin, and mitomycin on day 36.

After 1 week of rest, patients in all regimens receive a second 4-week course of systemic chemotherapy.

Cohorts of 3-10 patients are sequentially enrolled until the maximum tolerated dose (MTD) of chemotherapy and chemoembolization is determined. The MTD is defined as the dose preceding that at which at least 4 of 10 patients experience dose-limiting toxicity.

* Phase III: Patients are stratified according to liver volume involvement (less than 25% vs 25-50% vs more than 50% to less than 75%) and participating center. Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive irinotecan IV over 60-90 minutes, leucovorin calcium IV, and fluorouracil IV over 10 minutes on days 1, 8, 15, and 22. Courses repeat every 6 weeks in the absence of disease progression.
  * Arm II: Patients receive chemotherapy as in arm I. Patients undergo hepatic chemoembolization with cisplatin, doxorubicin, and mitomycin on day 36. Chemotherapy repeats every 6 weeks in the absence of disease progression. Chemoembolization may repeat every 6 weeks for 2-4 courses as necessary.

Patients in phase III are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 9-18 patients will be accrued for phase I of this study. (Phase I closed to accrual as of 10/14/02.) Approximately 315 patients will be accrued for phase III of this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic colorectal adenocarcinoma

  * Measurable metastasis to liver at least 1.0 cm

    * Less than 75% of total liver volume
  * Known extrahepatic disease limited to lymph nodes and less than 2 cm
  * No ascites
* Ineligible for surgery

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 2,000/mm^3
* Platelet count at least 90,000/mm^3
* No bleeding diathesis not correctable by standard therapy

Hepatic:

* Ineligible if all of the following criteria are concurrently present:

  * High risk of hepatic failure (more than 50% liver involvement by tumor)
  * Bilirubin greater than 2.0 mg/dL
  * SGOT greater than 100 U/L
  * Lactate dehydrogenase greater than 425 U/L
* No hepatic encephalopathy
* No portal vein occlusion without hepatopedal collateral flow demonstrated by angiography
* No portal hypertension with hepatofugal flow

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No myocardial infarction within the past 6 months
* No evidence of congestive heart failure
* No severe peripheral vascular disease that would preclude catheterization

Other:

* No severe allergy or intolerance to contrast media, narcotics, sedatives, or atropine
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No more than 1 prior adjuvant immunotherapy regimen for colon cancer

Chemotherapy:

* At least 6 months since prior adjuvant chemotherapy and recovered
* No more than 1 prior adjuvant chemotherapy regimen for colon cancer
* No prior hepatic arterial infusion chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 1 month since prior radiotherapy
* No prior hepatic radiotherapy

Surgery:

* At least 1 month since prior surgery
* Prior surgical resection or ablation of liver metastases allowed

Other:

* No other concurrent therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-11-01 (Actual); Primary Completion 2002-09-25 (Actual); Study Completion 2002-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C. Soulen, MD, Study Chair — Abramson Cancer Center at Penn Medicine
Locations (9):
- United States (9):
  - Arizona Cancer Center, Tucson, Arizona
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Texas - MD Anderson Cancer Center, Houston, Texas